CLINICAL TRIAL: NCT00721656
Title: A Randomized, Double Blind, Placebo Controlled, Phase 2 Study of KLS-0611 in Patients With Dry Eye Syndromes
Brief Title: Phase 2 Study of KLS-0611 in Patients With Dry Eye Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KLS1201
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes; Corneal diseases; Conjunctival Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases; Conjunctival Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KLS-0611 (Experimental)
  Interventions: Drug: KLS-0611

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: KLS-0611
  Arms: KLS-0611

SUMMARY:
To evaluate the efficacy and safety of KLS-0611 compared to placebo in patients with dry eye syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Corneal and conjunctival damage
* Insufficiency of lacrimal secretion
* Ocular symptom

Exclusion Criteria:

* Severe ophthalmic disorder
* Punctual plugs or surgery for occlusion of the lacrimal puncta

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)

PRIMARY OUTCOMES:
Corneal-conjunctival staining | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Japan, Hokkaido Region
  - Japan, Kansai Region
  - Japan, Kanto Region
  - Japan, Kyushu Region
  - Japan, Shikoku Region